CLINICAL TRIAL: NCT03892603
Title: Rotator Cuff Related Shoulder Pain: Does The Type of Exercise Influence Outcome? - A Randomized Controlled Trial
Brief Title: Does The Type of Exercise Influence Outcome in Rotator Cuff Related Shoulder Pain
Acronym: RCT-RCRSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Associate Professor, Faculty of Medicine, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT RCRSP 2019
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Shoulder Pain; Rotator Cuff Injury; Rotator Cuff Tendinitis; Rotator Cuff Impingement Syndrome
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries; Shoulder Impingement Syndrome | interventions — Educational Status; Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strengthening exercises program (Experimental)
  Interventions: Other: Strengthening exercises program
- Motor control exercises program (Experimental)
  Interventions: Other: Motor control exercises program
- Education and advice (Active Comparator)
  Interventions: Other: Education and advice

INTERVENTIONS:
Other: Strengthening exercises program — Participants from this group will be given a progressive shoulder strengthening exercises program based on 1 RM that will involve isometric, concentric and eccentric contractions. The exercises will target shoulder internal/external rotators and abductors and the scapular muscles. They will have to exercise every other day for 12 weeks. At each session with the therapist (6 over a 12 week period), strength will be reassessed and the program will be progressed accordingly. Any questions or concerns will also be addressed and participants will be requested to complete a paper based or digital record of their exercise participation.
  Arms: Strengthening exercises program
Other: Motor control exercises program — Each session will start with a series of clinical tests that will look at the influence of different corrections to alleviate symptoms during upper limb movements.The tests will be performed in a sequential format through four key areas: thoracic repositioning, scapula facilitation, humeral head procedures and neuromodulatory techniques. If a correction reduces pain, that technique will then be performed as exercises and incorporated into the participant's functional movement. In addition, motor control exercises during arm elevation, progressed through a standardized 6-phase retraining sequence, will be executed. Retraining phases will be graded according to: 1) resistance applied on the shoulder; and 2) use or non-use of feedback. Once participants reach pain free execution, the program will be progressed into re-education exercises according to the participants' work, sport and activities of daily living and will incorporate activities involving the upper and lower limbs.
  Arms: Motor control exercises program
Other: Education and advice — Each participant will be given written information about the shoulder (anatomy and function), basic pain science and will be directed to the Internet to watch a series of carefully selected educational videos. Comprehensive written advice will include: Information about the shoulder and the condition; Pain neuroscience; Activity modification (when to increase and decrease); Pain management (night and day); A series of educational videos to watch with 2 questions to answer per video: a) what was the most important message? and b) was there anything you didn't understand in the video?
  Arms: Education and advice

SUMMARY:
Rotator cuff related shoulder pain (RCRSP) is the most common shoulder disorder and its chronicization leads to multiple consequences such as early retirement, absenteeism from work, decreased participation and quality of life and expensive yearly healthcare costs (128 739 687 $ according to CNESST). Even though scientific evidence has shown that prioritising physiotherapy exercises over surgery for the initial management of RCRSP is a great way to save on healthcare costs without compromising quality, it does not always result in a resolution of symptoms and patients' quality of life can still be affected thereafter: up to 30% of people with RCRSP remain symptomatic despite rehabilitation interventions. This lack of therapeutic success could be explained by a multitude of factors, but a central issue that can explain a lack of improvement is an inappropriate dosage or choice of exercises prescribed. The purpose of this study is to compare the effectiveness of 3 non-operative methods of delivering shoulder management (2 types of exercises and an advice and education only group) on symptoms and functional limitations for people with RCRSP. Results from this project should help us further our knowledge on which non-operative treatment to promote with patients presenting with RCRSP, thus decreasing the proportion of individuals experiencing pain even after going through a rehabilitation program.

DETAILED DESCRIPTION:
Context : Musculoskeletal injuries lead to the second largest number of years lived with a disability, just behind mental health problems. Among those, shoulder problems are widespread and become even more common over the years. 70% of the population will experience an episode of shoulder pain during their lifetime and 30% of people over 65 years old live with daily shoulder pain. Unfortunately, the resolution of shoulder pain is often slow and incomplete and about 40 to 50% of symptomatic individuals will still experience pain one year after the onset of their painful episode. Rotator cuff related shoulder pain (RCRSP) is the most common type of injury in this region. This is a broad term that includes subacromial conflict syndrome, rotator cuff tendinopathy, and non-traumatic tears of rotator cuff tendons. There is ample evidence to suggest that physiotherapy exercises are the preferred approach as the first intervention for managing this condition, without having an impact on the quality of recovery. Unfortunately, for many patients, this approach does not lead to a significant decrease in symptoms and may result in a decrease in their quality of life. This lack of therapeutic success could be explained by a multitude of factors: psychosocial, physical, genetic, lifestyle, complex problems related to pain and lack of adherence to the exercise program. Another important element that may explain this lack of improvement is an inappropriate dosage and / or choice of prescribed exercises.

Objectives : The primary objective of this randomized clinical trial is to compare the short, medium, and long-term effects, in terms of symptoms and functional limitations, of three different options (education, strengthening, motor control) for the management of individuals with RCRSP. A secondary objective is to explore the effects of these interventions on shoulder control (acromiohumeral distance), subacromial structures (thickness of the supraspinatus and infraspinatus tendons), kinesiophobia and pain catastrophization.

Methods : 123 individuals between the ages of 18 and 75 with RCRSP for more than 3 months will be recruited and randomly assigned to one of three 12-week interventions: 1) counseling and education only; 2) scapulohumeral and scapulothoracic muscles strengthening exercises; 3) Motor control program paired with global exercises. Before being assigned to their respective group, patients will undergo an initial assessment including self-administered questionnaires on symptoms and functional limitations (QuickDASH, WORC, BPI-SF, TSK, PCS) as well as ultrasound measurements of the shoulder (acromiohumeral distance and thickness of supraspinatus and infraspinatus tendons). The questionnaires will be administered again at 3, 6, 12 and 24 weeks after the inclusion of the participants in the project and the ultrasound measurements will be re-evaluated at 12 weeks. Initial demographic data will be compared (independent t-test and square-test) to establish comparability of groups. Two-way ANOVA analyzes will be used to analyze and compare the effects of the three programs on the primary outcome (QuickDASH) and the other questionnaires (3 interventions x 5 times [0, 3, 6, 12 and 24 weeks]) as well as for the ultrasound measurements (3 interventions X 2 times [0 and 12 weeks]) (SPSS 25, proc GENLIN).

Expected results : The hypothesis is that the two exercises groups will show better results in terms of symptoms and functional limitations compared to the group consisting solely of counseling and education. The motor control program should allow a faster improvement of symptoms and functional limitations than the reinforcement program because, by improving muscular recruitment patterns and scapular kinematics, it will reduce control deficits and thus the probabilities to feel pain. Finally, all groups should show a decrease in kinesiophobia and pain catastrophization, but the exercises groups should result in a larger one, as participants will have to move their arms in ranges previously limited by pain and / or fears related to pain, or perform muscle contractions of near maximal intensity.

ELIGIBILITY:
Inclusion Criteria:

* Pain of at least 3 months duration
* At least one positive response in the three following categories

  1. Painful arc of movement (flexion; abduction)
  2. Positive shoulder impingement test (Neer; Kennedy-Hawkins)
  3. Pain during resisted isometric shoulder contraction (external rotation; abduction; Jobe)

Exclusion Criteria:

* Clinical signs of massive rotator cuff tears (gross weakness of rotator cuff muscles in the absence of pain)
* Other shoulder disorders (arthritis, adhesive capsulitis, fracture, acromioclavicular joint pathology)
* Undergone previous shoulder surgery on the same side
* Presence of significant co-morbidity (neurological disorders, rheumatoid arthritis)
* Symptomatic cervical spine pathology defined as reproduction of symptoms with active physiological cervical spine movement
* Inability to understand French or English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
Change in symptoms and functional limitations from baseline to 3 weeks: QuickDASH | 0 and 3 weeks
  The QuickDASH is a self-reported questionnaire that includes 11 items measuring physical disability and symptoms. This tool uses a 5-point (1-5) Likert scale. The total out of 55 is then reported to a score from 0 to 100. Score ranges from 0 (no disability) to 100 (most severe disability).
Change in symptoms and functional limitations from baseline to 6 weeks: QuickDASH | 0 and 6 weeks
  The QuickDASH is a self-reported questionnaire that includes 11 items measuring physical disability and symptoms. This tool uses a 5-point (1-5) Likert scale. The total out of 55 is then reported to a score from 0 to 100. Score ranges from 0 (no disability) to 100 (most severe disability).
Change in symptoms and functional limitations from baseline to 12 weeks: QuickDASH | 0 and 12 weeks
  The QuickDASH is a self-reported questionnaire that includes 11 items measuring physical disability and symptoms. This tool uses a 5-point (1-5) Likert scale. The total out of 55 is then reported to a score from 0 to 100. Score ranges from 0 (no disability) to 100 (most severe disability).
Change in symptoms and functional limitations from baseline to 24 weeks: QuickDASH | 0 and 24 weeks
  The QuickDASH is a self-reported questionnaire that includes 11 items measuring physical disability and symptoms. This tool uses a 5-point (1-5) Likert scale. The total out of 55 is then reported to a score from 0 to 100. Score ranges from 0 (no disability) to 100 (most severe disability).

SECONDARY OUTCOMES:
Change in symptoms and functional limitations from baseline to 3 weeks: WORC (Western Ontario Rotator Cuff Index) | 0 and 3 weeks
  The WORC index is a disease-specific questionnaire developed to measure health related quality-of-life of individuals suffering from RC disorders. It contains 21 items divided into five sections: physical symptoms, sports/recreation, work, lifestyle and emotions. Each question uses a visual analogue scale representing a 100 point scale (0-100). Maximum score is 2100 and minimum is 0. Total score is reported as a percentage where 0% represents lowest functional status level and 100% represents the highest level.
Change in symptoms and functional limitations from baseline to 6 weeks: WORC | 0 and 6 weeks
  The WORC index is a disease-specific questionnaire developed to measure health related quality-of-life of individuals suffering from RC disorders. It contains 21 items divided into five sections: physical symptoms, sports/recreation, work, lifestyle and emotions. Each question uses a visual analogue scale representing a 100 point scale (0-100). Maximum score is 2100 and minimum is 0. Total score is reported as a percentage where 0% represents lowest functional status level and 100% represents the highest level.
Change in symptoms and functional limitations from baseline to 12 weeks: WORC | 0 and 12 weeks
  The WORC index is a disease-specific questionnaire developed to measure health related quality-of-life of individuals suffering from RC disorders. It contains 21 items divided into five sections: physical symptoms, sports/recreation, work, lifestyle and emotions. Each question uses a visual analogue scale representing a 100 point scale (0-100). Maximum score is 2100 and minimum is 0. Total score is reported as a percentage where 0% represents lowest functional status level and 100% represents the highest level.
Change in symptoms and functional limitations from baseline to 24 weeks: WORC | 0 and 24 weeks
  The WORC index is a disease-specific questionnaire developed to measure health related quality-of-life of individuals suffering from RC disorders. It contains 21 items divided into five sections: physical symptoms, sports/recreation, work, lifestyle and emotions. Each question uses a visual analogue scale representing a 100 point scale (0-100). Maximum score is 2100 and minimum is 0. Total score is reported as a percentage where 0% represents lowest functional status level and 100% represents the highest level.
Change in pain from baseline to 3 weeks: BPI-SF (Brief Pain Inventory-Short Form) | 0 and 3 weeks
  The BPI-SF is a validated 9 item self-administred questionnaire used to assess the intensity of pain and the interference of the pain on the patient's life. Each item is scored on a 10-point Likert scale.
Change in pain from baseline to 6 weeks: BPI-SF | 0 and 6 weeks
  The BPI-SF is a validated 9 item self-administered questionnaire used to assess the intensity of pain and the interference of the pain on the patient's life. Each item is scored on a 10-point Likert scale.
Change in pain from baseline to 12 weeks: BPI-SF | 0 and 12 weeks
  The BPI-SF is a validated 9 item self-administered questionnaire used to assess the intensity of pain and the interference of the pain on the patient's life. Each item is scored on a 10-point Likert scale.
Change in pain from baseline to 24 weeks: BPI-SF | 0 and 24 weeks
  The BPI-SF is a validated 9 item self-administered questionnaire used to assess the intensity of pain and the interference of the pain on the patient's life. Each item is scored on a 10-point Likert scale.
Change in kinesiophobia from baseline to 3 weeks: TSK (Tampa Scale of Kinesiophobia) | 0 and 3 weeks
  The Tampa Scale of Kinesiophobia (TSK) is a 17 item self-administered questionnaire that measures beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging and painful movements should be avoided. It uses a 4-point Likert scale and total score ranges from 17 (lowest degree of kinesiophobia) to 68 (highest degree of kinesiophobia).
Change in kinesiophobia from baseline to 6 weeks: TSK (Tampa Scale of Kinesiophobia) | 0 and 6 weeks
  The Tampa Scale of Kinesiophobia (TSK) is a 17 item self-administered questionnaire that measures beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging and painful movements should be avoided. It uses a 4-point Likert scale and total score ranges from 17 (lowest degree of kinesiophobia) to 68 (highest degree of kinesiophobia).
Change in kinesiophobia from baseline to 12 weeks: TSK (Tampa Scale of Kinesiophobia) | 0 and 12 weeks
  The Tampa Scale of Kinesiophobia (TSK) is a 17 item self-administered questionnaire that measures beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging and painful movements should be avoided. It uses a 4-point Likert scale and total score ranges from 17 (lowest degree of kinesiophobia) to 68 (highest degree of kinesiophobia).
Change in kinesiophobia from baseline to 24 weeks: TSK (Tampa Scale of Kinesiophobia) | 0 and 24 weeks
  The Tampa Scale of Kinesiophobia (TSK) is a 17 item self-administered questionnaire that measures beliefs and behaviours related with pain, specially focusing on beliefs that pain is damaging and painful movements should be avoided. It uses a 4-point Likert scale and total score ranges from 17 (lowest degree of kinesiophobia) to 68 (highest degree of kinesiophobia).
Change in pain catastrophization from baseline to 3 weeks: PCS (Pain Catastrophizing Scale) | 0 and 3 weeks
  The Pain Catastrophizing Scale (PCS) is a 13 item self-administered questionnaire measuring the range of catastrophic thoughts and feelings (magnified threat, ruminating thoughts and feelings of helplessness) associated with pain that individuals may experience. Items are scored on a scale from 0 (not at all) to 4 (all the time). Total score ranges from 0 (minimum) to 52 (maximum).
Change in pain catastrophization from baseline to 6 weeks: PCS (Pain Catastrophizing Scale) | 0 and 6 weeks
  The Pain Catastrophizing Scale (PCS) is a 13 item self-administered questionnaire measuring the range of catastrophic thoughts and feelings (magnified threat, ruminating thoughts and feelings of helplessness) associated with pain that individuals may experience. Items are scored on a scale from 0 (not at all) to 4 (all the time). Total score ranges from 0 (minimum) to 52 (maximum).
Change in pain catastrophization from baseline to 12 weeks: PCS (Pain Catastrophizing Scale) | 0 and 12 weeks
  The Pain Catastrophizing Scale (PCS) is a 13 item self-administered questionnaire measuring the range of catastrophic thoughts and feelings (magnified threat, ruminating thoughts and feelings of helplessness) associated with pain that individuals may experience. Items are scored on a scale from 0 (not at all) to 4 (all the time). Total score ranges from 0 (minimum) to 52 (maximum).
Change in pain catastrophization from baseline to 24 weeks: PCS (Pain Catastrophizing Scale) | 0 and 24 weeks
  The Pain Catastrophizing Scale (PCS) is a 13 item self-administered questionnaire measuring the range of catastrophic thoughts and feelings (magnified threat, ruminating thoughts and feelings of helplessness) associated with pain that individuals may experience. Items are scored on a scale from 0 (not at all) to 4 (all the time). Total score ranges from 0 (minimum) to 52 (maximum).
Change in ultrasonographic measurement of acromiohumeral distance from baseline to 12 weeks | 0 and 12 weeks
  US images of AHD will be obtained with the participants seated in a standardized position with the arm at rest and at 60° of active abduction. US measures will be obtained by placing the transducer on the anterior aspect of the lateral surface of acromion along the longitudinal axis of the humerus in a frontal plane. The AHD will be measured using the build-in electronic caliper option by manually locating the superior aspect of the humeral head and the inferior aspect of acromion and then measuring the shortest linear distance between those two landmarks. For each upper limb position, three measurements will be taken.
Change in ultrasonographic measurement of supraspinatus tendon thickness from baseline to 12 weeks | 0 and 12 weeks
  Thickness of the supraspinatus (SS) tendon will be obtained with the medial aspect of the wrist against the ipsilateral anterior superior iliac spine. Measures will be obtained with the transducer perpendicularly, one centimeter behind to the anterolateral aspect of the surface of the acromion. The thickness of the SS tendon borders will be defined inferiorly as the first hyperechoic region above the anechoic articular cartilage of the humeral head, and the hyperechoic superior border of the tendon before the anechoic subdeltoid bursa.
Change in ultrasonographic measurement of infraspinatus tendon thickness from baseline to 12 weeks | 0 and 12 weeks
  Infraspinatus tendon thickness will be measured at the level of the posterior border of the acromion with the hand placed on the opposite shoulder.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Sébastien Roy, PT, PhD, Study Director — Laval University, Quebec, Qc (Canada)
Locations (1):
- Centre interdisciplinaire de recherche en réadaptation et intégration sociale (CIRRIS), Québec, Quebec, Canada

REFERENCES:
- [Derived] Dube MO, Desmeules F, Lewis JS, Roy JS. Does the addition of motor control or strengthening exercises to education result in better outcomes for rotator cuff-related shoulder pain? A multiarm randomised controlled trial. Br J Sports Med. 2023 Apr;57(8):457-463. doi: 10.1136/bjsports-2021-105027. Epub 2023 Feb 16. PMID 36796859
- [Derived] Dube MO, Desmeules F, Lewis J, Roy JS. Rotator cuff-related shoulder pain: does the type of exercise influence the outcomes? Protocol of a randomised controlled trial. BMJ Open. 2020 Nov 5;10(11):e039976. doi: 10.1136/bmjopen-2020-039976. PMID 33154058